CLINICAL TRIAL: NCT07084831
Title: A Prospective, Open-label, Single-arm, Multicenter Study Evaluating the Efficacy of One Year Treatment With Xanomeline/Trospium on Cognitive Impairment in Clinically Stable Adult Participants With Schizophrenia.
Acronym: SHINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Group for Research In Schizophrenia (Other)
Collaborators: Bristol-Myers Squibb (Industry); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-523060-20-00
Record Dates: First submitted 2025-07-23; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Psychosis; Cognitive Impairment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Intervention Model Description: Drug: Xanomeline/trospium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xanomeline/trospium (Experimental): Xanomeline/trospium that is provided to all participants
  Interventions: Drug: Xanomeline/trospium

INTERVENTIONS:
Drug: Xanomeline/trospium — Participants will receive xanomeline/trospium during the trial
  Other Names: KarXT/Cobenfy

SUMMARY:
Schizophrenia is a chronic, severe psychiatric disorder affecting approximately 1% of the global population. Symptoms are usually treated with antipsychotics (AP). All currently available APs work by blocking dopamine receptors in the brain. This is effective to treat the symptoms, but also leads to side-effects. Side effects contribute to poor medication adherence, resulting in frequent relapses and hospitalizations. In addition, the cognitive symptoms are not treated by the current APs.

Xanomeline/Trospium (US brand name: COBENFY™) is a novel combination of xanomeline tartrate (a muscarinic agonist) and trospium chloride (a muscarinic antagonist). It offers significant therapeutic benefits through its unique mechanism of action, selectively targeting central muscarinic acetylcholine receptors while mitigating peripheral side effects. This makes Xanomeline/Trospium a promising alternative to existing antipsychotics. This combination has demonstrated robust efficacy in reducing psychotic symptoms in recent trials, with a favorable side-effect profile. These findings led to the FDA approval of Xanomeline/Trospium (Cobenfy) in 2024 for the treatment of schizophrenia. Preliminary exploratory cognitive assessments in these trials have suggested potential pro-cognitive effects, particularly in domains such as attention and working memory, although these were not powered to detect changes in cognition 1,2.

Most antipsychotic trials include only superficial cognitive assessments, often limited to brief screening tools or exploratory endpoints. Furthermore, few studies explore the longitudinal course of cognition over extended treatment periods. In the current study, we propose to conduct a deep-dive into cognitive functioning in patients with schizophrenia who are treated with Xanomeline/Trospium for a one-year period. Cognitive functioning is highly integrated within the study design with other relevant domains, such as clinical symptoms, functioning, and quality of life, offering a more holistic picture of treatment impact. By focusing on cognition as a primary outcome in a naturalistic yet rigorous study design, this trial addresses a critical unmet need in schizophrenia research and has the potential to inform a paradigm shift in treatment strategies beyond symptom stabilization toward cognitive and functional recovery. By investing in this level of cognitive phenotyping, the study aligns with calls from both scientific and regulatory bodies for precision in cognitive outcomes and contributes to a growing body of work aimed at establishing cognition as a co-primary treatment target in schizophrenia.

DETAILED DESCRIPTION:
Design:

This is a phase III, prospective, open-label, single-arm, international, multicenter study. At visit 1, the informed consent is signed and screening is performed to confirm eligibility. At visit 2, baseline measures are performed, and the new treatment is initiated. Between visit 1 and 4 the current antipsychotic treatment is tapered down. At visit 3, 4, 5, 7 and 9 participants' general wellbeing and safety is assessed. At visit 6, 8 and 10, baseline measures are repeated. Between visit 6-7, visit 7-8, visit 8-9 and visit 9-10, a phone call is planned to assess general psychopathology, adverse events and concomitant medication. The treatment duration is one year for each participant; no additional follow-up is planned. All participants are treated with Xanomeline/Trospium open label.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 55 years of age.
2. Be willing and able to provide informed consent, after the nature of the study has been fully explained.
3. Have a current DSM-5 diagnosis of schizophrenia, schizoaffective order or schizophreniform disorder, which needs to be confirmed by MINI.
4. Have all PANSS positive items + G8 and G10 ≤4 at screening.
5. Be on a stable dose of any second generation antipsychotic drug (in monotherapy) prescribed to treat psychosis, for at least 4 weeks prior to the screening visit.
6. Have a SCIP total below 70.
7. Test negative for pregnancy at the screening visit and must be using a dual method contraceptive method during the study and 30 days after the study, if being a female of childbearing potential

Exclusion Criteria:

1. Be pregnant or breast-feeding, in case of female participant.
2. Be at significant risk of committing suicide. This is defined as: participants with active suicidal ideation with some intent to act, without specific plan ("Yes" to question 4 of the Columbia-Suicide Severity Rating Scale (C-SSRS)) or active suicidal ideation with specific plan and intent ("Yes" to question 5 of the C-SSRS), followed by an assessment by the treating clinician who determines it is not safe for the participant to participate in the study .
3. Currently meet DSM-5 criteria for a manic episode or major depressive disorder as confirmed by the MINI.
4. Currently meeting DSM-5 criteria for severe substance and/or alcohol use disorder as confirmed by the MINI (≥6 on module K for alcohol use disorder and/or ≥6 on module J for substance use disorder, unless being in early or sustained remission).

   A positive urine toxicology for phencyclidine, amphetamines, opiates (unless participant has a valid prescription for short-term use), cocaine, or alcohol (clinically significant alcohol use in the opinion of the Investigator). Nicotine and caffeine use is allowed. Stimulants and cannabis is allowed when used sporadically and recreationally as per the judgement of the clinician.
5. Present with intellectual disability, drug-induced psychosis, or history of clinically significant brain trauma as per the judgement of the clinician.
6. Have urinary retention, moderate or severe hepatic impairment, gastric retention, history of hypersensitivity to Xanomeline/Trospium or trospium chloride, untreated narrow-angle glaucoma, or any other medical condition (as per the participant's medical files) that makes, as per the judgement of the clinician, the patient unsuitable for the study.
7. Currently use clozapine, a long-acting injectable antipsychotic, or anticholinergic treatment*.
8. Expect to require more than the allowed psychotropic concomitant medication during the study (from baseline on). This is defined as: needing benzodiazepines of more than 2 mg lorazepam equivalent (daily), quetiapine, antidepressants, mood stabilizers or benzodiazepines at a dose exceeding the allowed threshold. If these treatments are used at the screening visit, they must be tapered down before the baseline visit.
9. An eGFR of < 60 mL/min
10. Elevations in hepatic transaminases at screening ≥ 3× ULN for ALT and AST and/or bilirubin > 3 × ULN, unless in the context of Gilbert's syndrome.

    Note: Gilbert syndrome is an inherited disorder characterized by mild elevation of unconjugated bilirubin in the absence of hemolysis or other cause.
11. History of unstable hypertension or tachycardia as evidenced by:

    Blood pressure of ≥ 160/100 mmHg at screening and/or a heart rate of ≥ 110 bpm at screening
12. Clinically significant abnormal finding on the physical examination, medical history, ECG (at screening), or clinically significant laboratory results at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance after 24 weeks of treatment, relative to baseline. | 24 weeks
  The within-participant change in the BACS composite cognitive score from baseline to follow-up after 24 weeks.

SECONDARY OUTCOMES:
Change in negative symptoms after 12 weeks and 24 weeks of treatment, relative to baseline. | 12 and 24 weeks
  The within-participant change in the PANSS negative subscale from baseline to follow-up after 12 weeks and 24 weeks.
Change in FUNSAT scores for ATM banking, ticket kiosk, and medication management after 24 weeks of treatment, relative to baseline | 24 weeks
  The within-participant change in the FUNSAT scores for ATM banking, ticket kiosk and medication management from baseline to follow-up after 24 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- Sheba Medical Center, Ramat Gan, Israel
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Group data can be requested.